CLINICAL TRIAL: NCT04620031
Title: A Multi-Center, Randomized, Single-Blind, Propofol-Controlled Phase III Clinical Study Evaluating Sedation of Intravenous Administration of HSK3486 Injectable Emulsion in ICU Patients Undergoing Mechanical Ventilation
Brief Title: A Study Evaluating Sedation of Intravenous Administration of HSK3486 Injectable Emulsion in ICU Patients Undergoing Mechanical Ventilation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSK3486-307
Record Dates: First submitted 2020-10-21; First posted 2020-11-06 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Sedation in Intensive Care
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): HSK3486 for Sedation
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): Propofol for Sedation
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — Loading Dose：0.1 mg/kg, infused with 4 min ± 30 s； Maintenance Dose：Maintenance is started at 0.3 mg/kg/h, and the dose can be adjusted up and down by 0.05-0.1 mg/kg/h. Range of maintenance dose: 0.06-0.8 mg/kg/h
  Arms: HSK3486
Drug: Propofol — Loading Dose：0.5 mg/kg, infused with 4 min ± 30 s
  Maintenance Dose：Maintenance is started at 1.5 mg/kg/h, and the dose can be adjusted up and down by 0.25-0.5 mg/kg/h. Range of maintenance dose:
  0.3-4 mg/kg/h
  Arms: Propofol

SUMMARY:
This is a multi-center, randomized, single-blind, propofol-controlled phase III clinical study. In this study, ICU patients undergoing mechanical ventilation are expected to be enrolled and will be randomly assigned to the HSK3486 group and the propofol group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who require tracheal intubation for mechanical ventilation are expected to require 6-24 h of sedation after randomization;
2. The target RASS for the required sedation of patients ranges from +1 to -2 points;
3. Aged ≥ 18 and < 80 years old, with no gender requirement;
4. 18 kg/m2 ≤ BMI ≤ 30 kg/m2;
5. The patients or their family members fully understand the objectives and significance of this study, and voluntarily participate in this clinical study and sign the informed consent form.

Exclusion Criteria:

1. Patients known to be allergic to eggs, soy products, opioids and their antidotes, and propofol; patient having contraindications to propofol, opioids and their antidotes;
2. Patients who have received sedation for more than 3 days in the ICU or in the general ward before being transferred to the ICU before signing informed consent form;
3. Patients having the following medical history or evidence of any of the following at screening, which may increase sedation/anesthesia risk:

   1. Cardiovascular system: New York Heart Association (NYHA) Class III and IV heart failure, Adams-stokes syndrome; acute coronary syndrome (ACS) that occurs within 6 months before screening; bradycardia requiring medication and/or heart rate ≤ 50 beats/min; a history of severe arrhythmia such as II-III degree atrioventricular block (excluding patients using pacemakers); acute and chronic myocarditis; patients who require vasoactive drugs to maintain a normal blood pressure;
   2. Patients with mental system disorders (such as schizophrenia, depression, etc.) and cognitive disorders; patients with a history of abuse of psychotropic drugs and anesthetics; patients with a history of alcohol abuse within 3 months prior to screening; patients with a history of drug abuse; patients with a history of long-term use of psychotropic drugs, etc.;
   3. Severe hepatic and renal insufficiency (liver function: refer to child-pugh grade C, the scale is shown in Appendix 6; renal function: glomerular filtration rate eGFR ≤ 30 mL/(min•1.73 m2) [eGFR is calculated using the Modification of Diet in Renal Disease (MDRD) equation: eGFR = 175 × serum creatinine (SCr)-1.234 × age-0.179 × 0.79 (females)]; patients undergoing dialysis;
   4. Grand mal epilepsy and convulsion; craniocerebral injury, intracranial hypertension, cerebral aneurysm; a Glasgow coma scale (GCS) of ≤ 12 points (see Appendix 4 for the scale); a SOFA scale of > 9 points (see Appendix 5 for the scale); patients with high paraplegia and general paralysis;
   5. Expected survival of ≤ 72 h.
4. Pregnant or lactating females; women or men of child-bearing potential who are unwilling to use contraception through the study; subjects who are planning pregnancy within 1 month after the study (including male subjects);
5. Have participated in any other clinical trials within 1 month prior to screening;
6. Other conditions that patients are judged by the investigator to be unsuitable for participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Success rate of sedation | Within 24 hours of administration
  1) The time period during which the RASS is in the range of +1 to -2 accounts for ≥ 70% of the total duration of study administration and 2) Remedial treatment is not used.

SECONDARY OUTCOMES:
Mean qualified rate of sedation | Within 24 hours of administration
  Defined as the percentage of time period during which the RASS is in the range of +1 to -2 relative to the total duration of study administration
Use of study drug | Within 24 hours of administration
  the loading doses of HSK3486 and propofol, mean maintenance dose and total dose per unit weight per hour of HSK3486 or propofol, and the number of dose modifications and the number of top up doses during the maintenance period
Dose of remedial drugs per unit weight | Within 24 hours of administration
  the mean dose per unit weight per hour of other sedatives used to maintain the target sedation (RASS within +1 to -2 points)
Time to extubation | Within 24 hours after administration
  the time from intubation (applicable to patients who undergoes intubation after entering the ICU)/ICU admission (applicable to patients with intubation before entering the ICU) to extubation or the time from drug discontinuation to extubation
Time to recovery | Within 24 hours after administration
  the time for the subject to recover from sedation to full recovery of consciousness (RASS ≥ 0) after discontinuation of drug administration
Incidence of adverse events | From day -1 to 24 hours after administration
  safety endpoits

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, China

REFERENCES:
- [Derived] Liu Y, Zuo L, Li X, Nie Y, Chen C, Liu N, Chen M, Wu J, Guan X. Early sedation using ciprofol for intensive care unit patients requiring mechanical ventilation: a pooled post-hoc analysis of data from phase 2 and phase 3 trials. Ann Intensive Care. 2024 Oct 26;14(1):164. doi: 10.1186/s13613-024-01390-3. PMID 39455495
- [Derived] Liu Y, Peng Z, Liu S, Yu X, Zhu D, Zhang L, Wen J, An Y, Zhan L, Wang X, Kang Y, Pan A, Yan J, Zhang L, Liu F, Zeng J, Lin Q, Sun R, Yu J, Wang H, Yao L, Chen C, Liu N, Nie Y, Lyu J, Wu K, Wu J, Liu X, Guan X. Efficacy and Safety of Ciprofol Sedation in ICU Patients Undergoing Mechanical Ventilation: A Multicenter, Single-Blind, Randomized, Noninferiority Trial. Crit Care Med. 2023 Oct 1;51(10):1318-1327. doi: 10.1097/CCM.0000000000005920. Epub 2023 Jun 5. PMID 37272947
- [Derived] Liu Y, Chen C, Liu N, Tong L, Nie Y, Wu J, Liu X, Gao W, Tang L, Guan X. Efficacy and Safety of Ciprofol Sedation in ICU Patients with Mechanical Ventilation: A Clinical Trial Study Protocol. Adv Ther. 2021 Oct;38(10):5412-5423. doi: 10.1007/s12325-021-01877-6. Epub 2021 Aug 21. PMID 34417990